CLINICAL TRIAL: NCT05004324
Title: A Two-stage, Multi-center, Randomized, Double-Blind, Placebo Controlled, Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of FURESTEM-AD Inj. for Moderate to Severe Chronic Atopic Dermatitis
Brief Title: Safety and Efficacy of FURESTEM-AD Inj. for Moderate to Severe Atopic Dermatitis (AD)
Acronym: smart(FURIN)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kang Stem Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K0106
Record Dates: First submitted 2021-07-04; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-07

CONDITIONS: Dermatitis, Atopic
Keywords: Atopic Dermatitis; AD; Stem cell; Furestem
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Furestem-AD Inj. (Experimental): Investigational product name: FURESTEM-AD® inj. 5.0 X 10^7 cells/1.5 mL
  baseline (0week) Experimental group will receive Investigational product (FURESTEM-AD® inj. 5.0 X 10^7 cells/1.5 mL).
  After 12 weeks, Experimental group will receive placebo.
  Interventions: Biological: FURESTEM-AD® inj. 5.0 X 10^7 cells/1.5 mL; Biological: Placebo
- Placebo (Placebo Comparator): Placebo
  baseline (0week) Placebo comparator group will receive placebo.
  After 12 weeks, Placebo comparator group will receive Investigational product (FURESTEM-AD® inj. 5.0 X 10^7 cells/1.5 mL).
  Interventions: Biological: FURESTEM-AD® inj. 5.0 X 10^7 cells/1.5 mL; Biological: Placebo

INTERVENTIONS:
Biological: FURESTEM-AD® inj. 5.0 X 10^7 cells/1.5 mL — the following study drug is injected respectively into both upper arms, both thighs, and abdomen (total of 5 regions)
Biological: Placebo — the following study drug is injected respectively into both upper arms, both thighs, and abdomen (total of 5 regions)

SUMMARY:
This clinical trial study is two-stage, multi-center, randomized, double-blind, placebo controlled, phase 3 clinical trial to evaluate the efficacy and safety of FURESTEM-AD Inj. for moderate to severe chronic atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 years and older at time of informed consent
2. Subjects diagnosed with atopic dermatitis based on the Hanifin and Rajka diagnostic criteria
3. Subjects with chronic atopic dermatitis that has been present for at least 1 year before screening
4. Subjects with moderate to severe atopic dermatitis as indicated by:

   * EASI score ≥ 16 points at the time of screening and baseline (Day 1),
   * IGA score ≥ 3 points at the time of screening and baseline (Day 1), and
   * BSA affected by atopic dermatitis ≥ 10% at the time of screening and baseline (Day 1)
5. Subjects who have documented history of insufficient response to stable use of atopic dermatitis treatment within 24 weeks before screening, or inability to receive such treatment because of safety issues
6. Subjects who are willing to apply a stable dose of non-medicated topical moisturizer at least twice daily for at least 7 days before the baseline (Day 1) visit and the duration of the study
7. Women of childbearing potential who use appropriate contraceptive methods during this trial period
8. Subjects who have voluntarily agreed to participate in this trial in writing

Exclusion Criteria:

1. Subjects with the following history of disease or surgery/procedure at screening

   1. Malignancy or lympho-proliferative disease within 5 years before screening (except completely treated carcinoma in situ of the cervix, or completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin)
   2. organ transplants
   3. History of mental illness, drug or alcohol abuse within 2 years before screening, as per Investigator's opinion
2. Subjects with the following underlying disease at screening

   1. Chronic active, acute infection or superficial skin infections requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals or antifungals;
   2. Skin diseases, pigmentation, or extensive scarring other than atopic dermatitis that may affect the efficacy evaluations of the study
3. Renal dysfunction with serum creatinine level > 2.0 mg/dL at screening
4. Liver dysfunction with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels exceeding 2.5 times the upper limit of the normal range (ULN) at the time of screening
5. Subjects with the history of using leukotriene receptor antagonists, systemic steroids, phototherapy, systemic immunosuppressants/modulators including janus kinase (JAK) inhibitors, and/or any other systemic therapy (not mentioned in Exclusion Criteria 6 and 8) to treat atopic dermatitis or symptoms of atopic dermatitis (approved or off-label use) within 4 weeks before baseline (Day 1)
6. Subjects with the history of using systemic or topical antihistamines, topical corticosteroids (TCS), topical calcineurin inhibitors (TCIs), or topical phosphodiesterase 4 (PDE4) inhibitors within 2 weeks before baseline (Day 1)
7. Allergen immunotherapy within 6 months before baseline (Day 1)
8. Subjects with the history of receipt of the following treatments before baseline (Day 1)

   1. B cell-depleting agents including rituximab within 6 months
   2. Other biologics including dupilumab within 5 half-lives (if known) or 12 weeks, whichever is longer
9. Subjects with regular use (more than two times per a week) of a tanning booth/parlor within 4 weeks before screening visit
10. Subjects with the history of a live (attenuated) vaccine injection within 12 weeks before baseline (Day 1) or the plan to inject a live (attenuated) vaccine within 24 weeks after randomization
11. Subjects who are deemed to require prohibited concomitant medications drug/therapy during the study period
12. Subjects with uncontrolled chronic disease that might require administration of oral corticosteroids such as uncontrolled and severe asthma
13. Pregnant/lactating women and men and women of childbearing potential who plan to become pregnant or who refuse to use appropriate contraceptive methods during the study period
14. Subjects with the history of receipt of any investigational products or devices from another clinical trial within 4 weeks or 5 half-lives (if known) pior to screening
15. Positive serology for hepatitis B or C, or for HIV
16. Subjects with prior use of FURESTEM-AD
17. Subjects with history of anaphylaxis
18. Subjects who are deemed to have difficulty in performing this study by the judgment of the Investigator and those with other medical findings that are unsuitable for participation in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2021-06-29 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
EASI(Eczema Area and Severity Index)-50 | 12 weeks
  Ratio of subject whose Eczema Area and Severity Index (EASI) decreased over 50% as contrasted with baseline value

SECONDARY OUTCOMES:
EASI(Eczema Area and Severity Index)-75 | 2,4,8,12 weeks
  Ratio of subjects whose Eczema Area and Severity Index (EASI) decreased over 75% as contrasted with baseline value
EASI(Eczema Area and Severity Index)-50 | 2,4,8 weeks
  Ratio of subjects whose Eczema Area and Severity Index (EASI) decreased over 50% as contrasted with baseline value
EASI(Eczema Area and Severity Index) index | 2,4,8,12 weeks
  Change and rate of change in Eczema Area and Severity Index (EASI) index as contrasted with baseline value
IGA(Investigator's Global Assessment) Score | 2,4,8,12 weeks
  Proportion of subjects who Investigator's Global Assessment (IGA) score 0 or 1 and at least 2 points reduction in IGA score as contrasted with baseline value
SCORAD(SCORing Atopic Dermatitis)-50 | 2,4,8,12 weeks
  Ratio of subjects whose SCORing Atopic Dermatitis (SCORAD) decreased over 50% as contrasted with baseline value
SCORAD(SCORing Atopic Dermatitis) index | 2,4,8,12 weeks
  Change and rate of change in SCORing Atopic Dermatitis (SCORAD) index as contrasted with baseline value
BSA(Body Surface Area) | 2,4,8,12 weeks
  Change and rate of change in Body Surface Area (BSA) as contrasted with baseline value
Worst daily Pruritus NRS(Numerical Rating Scale) | 2,4,8,12 weeks
  Rate of change in Worst daily Pruritus Numerical Rating Scale (NRS) as contrasted with baseline value
Average daily Pruritus NRS(Numerical Rating Scale) | 2,4,8,12 weeks
  Rate of change in Average daily Pruritus Numerical Rating Scale (NRS) as contrasted with baseline value
Worst daily Pruritus NRS(Numerical Rating Scale) - 4 points | 2,4,8,12 weeks
  Proportion of patients at least 4 points reduction in Worst daily Pruritus Numerical Rating Scale (NRS) as contrasted with baseline value
POEM(Patient-Oriented Eczema Measure) | 2,4,8,12 weeks
  Change and rate of change in Patient-Oriented Eczema Measure (POEM) as contrasted with baseline value
DLQI(Dermatology Life Quality Index) | 2,4,8,12 weeks
  Change and rate of change in Dermatology Life Quality Index (DLQI) as contrasted with baseline value
Rescue medicine | up to 12, 24 weeks
  Total number of use and consumed amount of rescue medicine

CONTACTS AND LOCATIONS:
Overall Officials: Yeonglib Park, professor (CI), Principal Investigator — Bucheon Hospital, Soonchunhyang University; Yangwon Lee, professor, Principal Investigator — Konkuk University Hospital; Sanguk Son, professor, Principal Investigator — Korea University; Bakrin Yoo, professor, Principal Investigator — Gangdong Kyunghee University Hospital; Jihyun Lee, professor, Principal Investigator — Seoul St. Mary's Hospital; Donghoon Lee, professor, Principal Investigator — Seoul National University Hospital; Chanho Na, professor, Principal Investigator — Chosun University Hospital; Yooin Bae, professor, Principal Investigator — Hallym University Dongtan Seongsim Hospital; Hyunchang Ko, professor, Principal Investigator — Yangsan Pusan National University Hospital; Younghyun Jang, professor, Principal Investigator — Kyungpook National University Hospital; Jeongeun Kim, professor, Principal Investigator — The Catholic University of Korea Eunpyeong St. Mary's Hospital; Minkyung Shin, professor, Principal Investigator — Kyunghee University Hospital; Sanghyun Cho, professor, Principal Investigator — Catholic University Incheon St. Mary's Hospital; Cheonuk Park, professor, Principal Investigator — Hallym University Gangnam Seongsim Hospital; Jooyeon Ko, professor, Principal Investigator — Hanyang University; Taeyoung Han, professor, Principal Investigator — Nowon Eulji University Hospital; Jiyoung Ahn, professor, Principal Investigator — National medical center
Locations (1):
- Chosun University Hospital, Gwangju, Jeollanam-do, South Korea

IPD SHARING:
Plan to Share IPD: No